CLINICAL TRIAL: NCT05212493
Title: The Effects of Medical Cannabis in Children With Autistic Spectrum Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Seach Sarid Ltd (Unknown); Canndoc Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0281-17-ASF; 20175083 (Registry Identifier: Israeli MOH)
Record Dates: First submitted 2021-12-12; First posted 2022-01-28 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Cannabis; co-morbid symptoms; ASD; Cannabidiol
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Seach CBD:THC 20:1 cannabis oil (Active Comparator): cannabis oil containing CBD:THC ratio of 20:1. plant material is grown by Seach LTD and oil manufactured by Nextar Pharma LTD.
  Interventions: Drug: Cannabis oil
- Candoc CBD:THC 20:1 cannabis oil (Active Comparator): cannabis oil containing CBD:THC ratio of 20:1. plant material is grown by Candoc LTD and oil manufactured by Panaxia LTD.
  Interventions: Drug: Cannabis oil

INTERVENTIONS:
Drug: Cannabis oil — Cannabis oil 20:1 CBD:THC ratio

SUMMARY:
Children with autism spectrum disorder (ASD) commonly exhibit comorbid symptoms such as aggression, hyperactivity and anxiety. Data on the effects of cannabidiol rich cannabis extract use for ASD is promising but still limited. The aim of this study is to investigate if oral cannabinoids treatment to children and young adults with ASD affect the comorbidities of autism, including sleep and eating problems, anxiety and violence.

The main objectives of the study are: 1) to characterize the effect of treatment with cannabis oil on comorbid symptoms of ASD; 2) to compare safety and efficacy of different cannabis products with identical CBD:THC ratio; 3) to investigate the effect of treatment on cognitive and adaptive behavior; and 4) to measure THC and CBD and metabolites levels in the blood of the patients.

In this study, patients diagnosed with ASD will be treated with cannabidiol-rich cannabis oil (CBD:THC ratio of 20:1). The researchers will collect parental reports on ASD comorbid symptoms before and bi-weekly during 6 months of the study period. Blood tests will be performed before and after three months of treatment. Blood tests include blood count, blood chemistry, hormones profile, phyto- and endo- cannabinoids and metabolites. Cognitive evaluation will be done before and after six months of treatment. Electroencephalogram (EEG) to exclude epilepsy will be performed before and after six months of treatment.

DETAILED DESCRIPTION:
Participants will be screened by the PI, a specialist neurologist. For those passing screening, license for Cannabis will be obtained at MOH.

Participants will pass tests such as ADOS (communication skills) and Wechsler (IQ), parents will fill questionnaires.

Treatment will start in a titration mode till improvement in some parameters is seen or till treatment failure decision is made.

Participants will be called for a check-up by mid-time (after 3 months) and their parents will fill questionnaires.

Participants will be called for a last check-up after 6 months from treatment beginning and pass again ADOS and Wechsler tests. Parents will fill questionnaires.

Secondary purposes of the trial:

To detect side-effects To assess treatment failure To assess treatment effect on sleep, motor restlessness and behavior. To examine treatment effect on hormonal profile

ELIGIBILITY:
Inclusion Criteria

* diagnosed with ASD by DSM
* IQ below 70. The investigator can include patients with IQ above 70 if they have significant ASD or comorbid symptoms.
* With significant behavior problems in for at least 6 months before recruitment

Exclusion Criteria:

* Epilepsy with clinical symptoms
* Current or previous treatment with cannabis
* Genetic disorder that can cause ASD symptoms
* Metabolic disorder
* immunologic disorder
* liver cancer
* Participants who, in the researcher's opinion, will not cooperate in the various research procedures
* Women which are pregnant or breastfeeding.
* Psychosis or schizophrenia or past or present schizoaffective disorder, in first-degree relatives
* History of substance abuse or abuse (including cannabis use disorder or alcohol addiction) in first-degree relatives
* Hypersensitivity to coconut oil / palm oil

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cannabinoids levels change | 3 months
  To compare CBD, THC their and metabolites blood levels before and after intervention
Changes in attention span | 6 months
  To characterize the effect of medical cannabis treatment on the attention span using Conners teacher questionnaires. Significant change is defined as a change of 10% in questionnaire score between baseline and 6 months.
Changes in cognitive level | 6 months
  To examine the effect of cannabis treatment on cognitive level using part of Wechsler test. Significant change is defined as a change of 10% in questionnaire score between baseline and 6 months.
Comparison of efficacy between two different cannabis oil products | 6 months
  To compare efficacy of medical cannabis products with the same CBD: THC ratio in terms of communication skills using ADOS test. Significant change is defined as a change of 10% in raw questionnaire score between baseline and 6 months.
Changes in adaptive behavior | 6 months
  To examine the effect of cannabis treatment on adaptive behavior as per ADOS test. Significant change is defined as a change of 10% in raw questionnaire score between baseline and 6 months.
Changes in violent behavior | 6 months
  To examine the effect of cannabis treatment on violent behavior as per specific trial-designed questionnaire. Significant change is defined as a change of 10% in questionnaire score between baseline and 6 months.

SECONDARY OUTCOMES:
Side effects | 6 months
  To identify side effects as per parents report in a specific trial-designed questionnaire. Significant change is defined as a change of 10% in new side effects as examined by questionnaire score between baseline and 6 months.
Therapeutic failure | 6 months
  To identify therapeutic failure reasons as per Professional expert opinion. Significant reason is defined as reason that will effect at least 20% of therapeutic failure cases.
Changes in sleep problems | 6 months
  To examine whether high concentration CBD cannabis oil is effective in improving sleep as per Sleep questionnaire. Significant change is defined as a change of 10% in raw questionnaire score between baseline and 6 months.
Changes in eating problems | 6 months
  To examine whether high concentration CBD cannabis oil is effective in improving eating as per eating questionnaire. Significant change is defined as a change of 10% in raw questionnaire score between baseline and 6 months.
Changes in hormonal profile | 3 months
  To compare hormonal profile measured as per by Hospital Lab SOP before and during treatment. measured hormones are: TSH, FT4, 17OH-testosterone, LH, prolactine. Significant change is defined as a clinically significant diversion from lab defined normal ranges, according to age and sex, between baseline and 3 months.
Changes in biochemical parameters | 3 months
  To compare liver enzymes measured as per by Hospital Lab SOP before and during treatment. Measured enzymes are: ALT, AST, GGT, Bilirubin. Significant change is defined as a clinicaly significant diversion (more than twice the Upper Limit of Noraml for each enzyme) from lab defined normal ranges, between baseline and 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Yes
the study protocol to be sahared upon request
Supporting Information: Study Protocol
Time Frame: during the duration of the trial
Access Criteria: for interested colleagues

REFERENCES:
- [Background] Iseger TA, Bossong MG. A systematic review of the antipsychotic properties of cannabidiol in humans. Schizophr Res. 2015 Mar;162(1-3):153-61. doi: 10.1016/j.schres.2015.01.033. Epub 2015 Feb 7. PMID 25667194
- [Background] Whiting PF, Wolff RF, Deshpande S, Di Nisio M, Duffy S, Hernandez AV, Keurentjes JC, Lang S, Misso K, Ryder S, Schmidlkofer S, Westwood M, Kleijnen J. Cannabinoids for Medical Use: A Systematic Review and Meta-analysis. JAMA. 2015 Jun 23-30;313(24):2456-73. doi: 10.1001/jama.2015.6358. PMID 26103030
- [Background] Barchel D, Stolar O, De-Haan T, Ziv-Baran T, Saban N, Fuchs DO, Koren G, Berkovitch M. Oral Cannabidiol Use in Children With Autism Spectrum Disorder to Treat Related Symptoms and Co-morbidities. Front Pharmacol. 2019 Jan 9;9:1521. doi: 10.3389/fphar.2018.01521. eCollection 2018. PMID 30687090

DOCUMENTS (1):
  • Study Protocol (2020-08-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT05212493/Prot_000.pdf